CLINICAL TRIAL: NCT03411018
Title: The Impact of Modifications on Respiratory Management of Preterm Infants on the Death or Bronchopulmonary Dysplasia Outcome
Brief Title: Respiratory Management of Preterm Infants and Bronchopulmonary Dysplasia
Status: Completed | Type: Observational
Sponsor: Manuel Sanchez Luna (Other)
Responsible Party: Sponsor-Investigator, Manuel Sanchez Luna, Head of Neonatology, Clinical Professor, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: CEIC 84/17
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: lung protective strategies; Less invasive respiratory support; preterm infant
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Conventional respiratory managed group.: Preterm infants born with less than 32 weeks gestational age (wGA) that entered in the neonatal Intensive care unit (NICU) from January 1 2012 to December 31 2013. These preterm infants were managed according to prior ventilatory protocol: Prophylactic Continuous positive airway pressure (CPAP) in delivery room, early surfactant administration by INSURE technique and volume target mechanical ventilation with rescue high frequency ventilation when needed. Mechanical ventilation exposure will be analyzed
  Interventions: Other: Mechanical ventilation exposure
- Less invasive managed group: Preterm Infants born with less than 32wGA that entered the NICU from January 1 2014 to December 31 2017. This infants are managed according to the actual ventilatory protocol. Prophylactic CPAP in delivery room, early surfactant administration by less invasive technique, nasal Synchronized positive pressure ventilation for CPAP failure and early rescue high frequency ventilation with minimally target volume.Mechanical ventilation exposure will be analyzed
  Interventions: Other: Mechanical ventilation exposure

INTERVENTIONS:
Other: Mechanical ventilation exposure

SUMMARY:
This observational study evaluates the impact of respiratory management modifications implemented in our institution on the intubation rates and the death or Bronchopulmonary Dysplasia (BPD) outcome.

DETAILED DESCRIPTION:
Less invasive respiratory management has been implemented in most neonatal units as well as lung protective ventilatory strategies when intubation is required in order to minimize ventilator induced lung injury.

In our institution a new ventilatory protocol including less invasive surfactant administration, Synchronized nasal positive pressure ventilation and early rescue High frequency ventilation has been implemented during 2013-14.

Hypothesis: New less invasive and lung protective strategies to prevent lung injury had been effective in reducing intubation rates.

ELIGIBILITY:
Inclusion Criteria:

All preterm Infants born with less than 32wGA admitted in our NICU.

Exclusion Criteria:

Congenital malformations and Known Chromosomal disorders,

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infant born with less than 32wGA since January 2012 to December 2017 admitted in our NICU.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
BRONCHOPULMONARY DySPLASIA | 36 weeks of postmenstrual age.
  Diagnosis of moderate-severe bronchopulmonary dysplasia (physiological definition)
mortality | before discharge
  death

SECONDARY OUTCOMES:
Mechanical ventilation | during hospitalization
  requirement of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ramos-Navarro, Principal Investigator — Gregorio Marañon, Hospital
Locations (1):
- Cristina Ramos-Navarro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No